CLINICAL TRIAL: NCT07152574
Title: ROTAO 1 - Feasibility and Safety of the TAVIPILOT Tele-operated Robot During Transcatheter Aortic Valve Replacement (TAVR/TAVI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caranx Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55005
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: TAVI(Transcatheter Aortic Valve Implantation)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of tele-operated TAVIPILOT Robot during the procedure (Experimental)
  Interventions: Device: TAVR using a tele-operated Robot

INTERVENTIONS:
Device: TAVR using a tele-operated Robot — TAVR procedure with TAVIPILOT tele-operated robot by Caranx Medical enhancing the precision of transcatheter aortic valve positioning during TAVR.

SUMMARY:
The TAVIPILOT tele-operated robot by Caranx Medical is an advanced intraoperative robotic assistance system designed to enhance the precision of transcatheter aortic valve positioning during TAVR. The system integrates with standard procedural workflows and enables remote manipulation of delivery system components, allowing for controlled, stable, and reproducible movements. TAVIPILOT facilitates accurate valve alignment and deployment, reducing operator variability. The robot is compatible with approved balloon-expandable transcatheter heart valves (Sapien 3 and Ultra, Edwards Lifesciences, USA) and standard catheterization lab infrastructure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥65
2. Indicated for transfemoral TAVR for severe aortic stenosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Investigational Device Safety | Periprocedural
  The primary objective is to evaluate investigational device-related safety, including the occurrence of investigational device-related conversion to open-heart surgery, investigational device-related valve embolization and investigational device-related trauma during progression through the ascending aorta and the native valve.
Investigational Device Safety | Periprocedural
  The investigational device-related safety will also be assessed by verifying the absence of major technical malfunctions.

SECONDARY OUTCOMES:
Device Usability | Periprocedural
  Evaluate clinical usability, assessed through customized questionnaires measuring clinician satisfaction, perceived ease of use, and integration of the devices into the procedural workflow.